CLINICAL TRIAL: NCT04159155
Title: Canadian Multi-arm Multi-stage Randomized Controlled Trial Assessing Front Line and Maintenance Treatment in Serous or p53 Mutant Endometrial Cancer
Brief Title: A Study of Various Treatments in Serous or p53 Abnormal Endometrial Cancer
Acronym: CAN-STAMP
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAN-STAMP; CAPCR 19-6178 (Other: Princess Margaret Cancer Centre)
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Carcinoma; P53 Mutation; Serous Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms; Cystadenocarcinoma, Serous | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Early Stage Cohort - Arm A (Experimental): Pelvic EBRT at 45Gy in 25 fractions, in 1.8Gy fractions daily, 5 days per week
  Interventions: Radiation: External Beam Radiation
- Early Stage Cohort - Arm B1 (Experimental): Vaginal high-dose rate brachytherapy 21 Gy in 3 fractions, prescribed to 5mm (i.e. 100% isodose at 5mm) from the cylinder/applicator surface and top along the upper third to half of the vagina (minimum 3cm, maximum 4cm).
  Interventions: Radiation: Vaginal high-dose rate brachytherapy
- Advanced Stage Cohort Arm C (Active Comparator): Observation
  Interventions: Other: Observation - no drugs
- Advanced Stage Cohort Arm D1 (Experimental): Investigational agent (niraparib), orally, at a dose of 200 mg, or 300 mg, once daily, based on baseline platelet count and weight.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Radiation: External Beam Radiation — Radiation therapy given outside the patient to a particular part of the body.
  Arms: Early Stage Cohort - Arm A
Drug: Niraparib — Oral drug
  Other Names: Zejula
  Arms: Advanced Stage Cohort Arm D1
Radiation: Vaginal high-dose rate brachytherapy — Internal radiation to the vagina
  Arms: Early Stage Cohort - Arm B1
Other: Observation - no drugs — Observation
  Arms: Advanced Stage Cohort Arm C

SUMMARY:
This is an umbrella, two-arm, multi-stage, phase II trial. The purpose of the trial in the early stage cohort is to determine if EBRT improves disease free survival (defined as the time from random assignment to disease recurrence or death from any cause) compared to vaginal brachytherapy after chemotherapy in women with serous or p53 aberrant endometrial cancer. The purpose of the trial in the advanced stage cohort is to determine if the maintenance with experimental treatment increases progression free survival, defined as the time from random assignment to disease progression or death from any cause.

DETAILED DESCRIPTION:
SC represents a rare and aggressive histologic subtype of endometrial cancer, associated with a poor prognosis. Moreover, there are marked molecular differences between EC and SC, showing the need to separate clinical trials to develop the personalized treatment paradigms that have improved outcomes in other tumor types, such as breast and lung cancer. Given the absence of consensus between pathologists on the diagnosis of SC, this trial will also incorporate a molecular marker, p53abd.

Several studies have been done in early stage endometrial cancer including diverse histologies, stages and molecular characteristics. Due to the heterogeneity of the patients, there is a lack of knowledge on the best treatment strategy. Even in cases where disease is apparently confined to the endometrium, the rate of recurrence is high. The role of radiation therapy in the management of this disease, with a high propensity for distant failures, remains elusive.

Furthermore, women with endometrial cancer often have multiple comorbidities, needing to optimize the treatment strategies and toxicities. It then results crucial to identify a strategy that is effective and results in limited toxicity.

Advanced or recurrent SC has a poor prognosis. There are no maintenance strategies currently approved for endometrial cancer and this is under investigation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pure serous endometrial carcinoma will be included. Other histotypes (endometrioid and clear cell) with abnormal/mutant-type p53 is acceptable.
* Local TP53 results must be available for Central review.
* Patients diagnosed with stage I, II tumors will be enrolled in the early stage cohort.
* Patients suitable for an optimal surgery.
* Eastern Cooperative Group (ECOG) performance status ≤ 2 (Karnofsky ≥60%).
* Life expectancy of greater than 3 months.
* Patients must have archival tissue available. If no tissue is available, tumor biopsy will be mandatory.
* Ability to understand and willing to sign a written informed consent document.
* Within 8 days of the proposed start of treatment, patients must have normal organ and marrow function.
* Women of child-bearing potential must agree to use effective contraceptive methods prior to study entry, during study participation, and for at least 30 days after the last administration of study medication.

Exclusion Criteria:

* Any other condition that would contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
* Mixed serous tumors without p53 aberration or with only subclonal p53 aberration
* Endometrial carcinosarcoma
* Patients being treated with radiotherapy within 4 weeks, or palliative radiotherapy encompassing >20% of the bone marrow within 1 week of starting study treatment.
* Patients who are receiving any other investigational agents.
* Participant has leptomeningeal disease, carcinomatous meningitis, symptomatic brain metastases, or radiologic signs of CNS hemorrhage. Note: Participants with asymptomatic brain metastases (i.e. off corticosteroids and anticonvulsants for at least 7 days) are permitted.
* Patients with evidence of fistula will be excluded.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study.
* Uncontrolled inter-current illness that would limit compliance with study requirements.
* Pregnant women are excluded.
* Known HIV-positive patients on antiretroviral therapy or active Hepatitis B or C are ineligible.
* Patients with a history of other malignancy ≤ 2 years prior to registration, with exceptions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival Rate | 3 years
  Time from random assignment until disease recurrence or death

SECONDARY OUTCOMES:
Overall Survival Rate | 5 years
  Time from enrollment until death.
Number Adverse Events Experienced | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No